CLINICAL TRIAL: NCT02264223
Title: The Effects of Processing and Matrices on Bioavailability of Red Clover Isoflavones in Healthy Women
Brief Title: The Bioavailability of Red Clover Isoflavones
Acronym: KLBIO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Southern Danish University (Unknown); Herrens Mark A/S (Unknown); Natur Drogeriet A/S (Unknown); Future Food Innovation (Industry)
Responsible Party: Principal Investigator, Per Bendix Jeppesen, Associate Prof., PhD, University of Aarhus
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: KLBIO 07-10-14
Record Dates: First submitted 2014-10-08; First posted 2014-10-15 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2015-12

CONDITIONS: Healthy
Keywords: Bioavailability; Isoflavones; Plasma; Human; Processing; Cross-over

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (5):
- Capsule (aglycone) (Active Comparator): single bolus 40mg isoflavone formulation of fermented extract in freeze-dried capsule.
  Fermented red clover isoflavones in aglycone form
  Interventions: Dietary Supplement: Fermented red clover isoflavones in aglycone form
- Tablet (aglycone) (Active Comparator): single bolus 40mg isoflavone aglycone formulation of fermented extract in freeze-dried tablet.
  Fermented red clover isoflavones in aglycone form
  Interventions: Dietary Supplement: Fermented red clover isoflavones in aglycone form
- Yoghurt (aglycone) (Active Comparator): single bolus 40mg isoflavone aglycone formulation of fermented extract mixed with yoghurt
  Fermented red clover isoflavones in aglycone form
  Interventions: Dietary Supplement: Fermented red clover isoflavones in aglycone form
- Liquid extract (aglycone) (Active Comparator): single bolus 40mg isoflavone aglycone formulation of fermented extract in liquid
  Fermented red clover isoflavones in aglycone form
  Interventions: Dietary Supplement: Fermented red clover isoflavones in aglycone form
- Tablet unfermented (glycoside) (Active Comparator): single bolus 40mg isoflavone aglycone equivalent tablet formulation of unfermented red clover isoflavones
  Unfermented glycosides (as aglycone equivalents)
  Interventions: Dietary Supplement: Unfermented glycosides (as aglycone equivalents)

INTERVENTIONS:
Dietary Supplement: Fermented red clover isoflavones in aglycone form — Fermented isoflavones in aglycone form
  Arms: Capsule (aglycone); Liquid extract (aglycone); Tablet (aglycone); Yoghurt (aglycone)
Dietary Supplement: Unfermented glycosides (as aglycone equivalents) — Unfermented aglycone equivalents in glycoside form
  Arms: Tablet unfermented (glycoside)

SUMMARY:
Previous literature has shown that the molecular form of isoflavones (as aglycones or glycosides) and food matrices can influence the bioavailability of these compounds in humans and hence their efficacy. To determine the effects of processing and food matrices on the bioavailability of active compounds derived from red clover the investigators will execute a 5 phase, cross-over design, open label, RCT using 20 healthy women aged between 18 to 40 years. Participants will receive 5 different formulations of red clover and bioavailability will be monitored in blood plasma using LC-MS.

DETAILED DESCRIPTION:
The aim of this study is to elucidate the effects food matrices and processing on the bioavailability of active compounds on the bioavailability of red clover derived isoflavones. 20 healthy participants will receive red clover derived isoflavones in five different formulations. The five formulations are split up into five phases:

Phase 1) Fermented extract in liquid form Phase 2) Fermented extract (freeze-dried) in capsule form Phase 3) Fermented extract (freeze-dried) in tablet form Phase 4) Fermented extract (concentrated) mixed in yogurt Phase 5) Un-fermented red clover in capsule or tablet form The trial will last 5-6 weeks for each participant. Plasma sample collection will take place both pre-and post- ingestion of a formulation, participants will receive blood tests at intervals -15 min, 0 min, 2hr, 4hr, 6hr, 8hr and 12hr (on the day of ingestion) and on the subsequent two mornings (24hr and 48hr) following the initiation of a phase. There will be a minimum. 5 day intervals between all phases (washout periods). Isoflavones biochanin A, formononetin, genistein and daidzein present in plasma will be detected using HPLC-MS for each phase, thus creating a bioavailability curve that can be compared to each of the other phases. The primary endpoint is to determine whether fermented extract is more bioavailable than unfermented extract.

ELIGIBILITY:
Inclusion criteria:

* Healthy women
* Age: 18-40 years

Exclusion Criteria:

* Habitual intake of soy products, chickpeas or other supplements with a high content of isoflavones
* Hormone therapy
* Pregnant or breastfeeding
* Taking drugs affecting uptake
* Participation in other clinical trials within the last 3 months
* Severe cardiovascular, psychiatric, neurological and / or kidney disease
* Alcohol or substance abuse
* Acute illness

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2014-10; Primary Completion 2022-05 (Actual); Study Completion 2022-05 (Actual)

PRIMARY OUTCOMES:
Bioavailability of isoflavones in terms of fermented vs unfermented formulations | -15min, 0hr, 2hr, 4hr, 6hr, 8hr, 12hr, 24hr, 48hr
  As measured by iAUC plasma concentrations of isoflavones over 48 hours

SECONDARY OUTCOMES:
Bioavailability of isoflavones in terms of matrices (tablet, capsule, yoghurt and liquid) | -15min, 0hr, 2hr, 4hr, 6hr, 8hr, 12hr, 24hr, 48hr
  As measured by iAUC plasma concentrations of isoflavones over 48 hours

CONTACTS AND LOCATIONS:
Overall Officials: Per B Jeppesen, Prof. PhD, Principal Investigator — University of Aarhus
Locations (1):
- Aarhus University Hospital, Aarhus, Central Jutland, Denmark